CLINICAL TRIAL: NCT02996825
Title: A Phase I Dose-Escalation Safety and Tolerability Study of MirvetuximabSoravtansine (IMGN853) and Gemcitabine in Patients With FRa-positive Recurrent Ovarian, Primary Peritoneal, Fallopian Tube, Endometrial Cancer, or Triple Negative Breast Cancer (TNBC)
Brief Title: Mirvetuximab Soravtansine and Gemcitabine Hydrochloride in Treating Patients With FRalpha-Positive Recurrent Ovarian, Primary Peritoneal, Fallopian Tube, Endometrial, or Triple Negative Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16294; NCI-2016-01913 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16294 (Other: City of Hope Medical Center)
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Recurrent Breast Carcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Recurrent Uterine Corpus Carcinoma; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms; Triple Negative Breast Neoplasms | interventions — Gemcitabine; mirvetuximab soravtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (IMGN853, gemcitabine hydrochloride) (Experimental): Patients receive mirvetuximab soravtansine IV on day 1 and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Cycles repeat every 3 weeks in the absence of disease progression or unexpected toxicity.
  Interventions: Drug: Gemcitabine; Drug: Gemcitabine Hydrochloride; Other: Laboratory Biomarker Analysis; Biological: Mirvetuximab Soravtansine; Other: Pharmacological Study

INTERVENTIONS:
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; FF 10832; FF-10832; FF10832; Gemcitabine HCI; Gemzar; LY-188011; LY188011
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Mirvetuximab Soravtansine — Given IV
  Other Names: IMGN853; M9346A-sulfo-SPDB-DM4
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of mirvetuximab soravtansine and gemcitabine hydrochloride in treating patients with folate receptor (FR) alpha-positive ovarian, primary peritoneal, fallopian tube, endometrial, or triple negative breast cancer that has come back. Mirvetuximab soravtansine is a monoclonal antibody, called mirvetuximab, linked to a chemotherapy drug called DM4. Mirvetuximab attaches to FOLR1 positive cancer cells in a targeted way and delivers DM4 to kill them. Drugs used in the chemotherapy, such as gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving mirvetuximab soravtansine and gemcitabine may work better in treating patients with FRalpha-positive ovarian, primary peritoneal, fallopian tube, endometrial, or triple negative breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of gemcitabine hydrochloride (gemcitabine) when given in combination with mirvetuximab soravtansine (IMGN853) to patients with FRalpha-positive recurrent ovarian, primary peritoneal, fallopian tube, endometrial cancer, or triple negative breast cancer (TNBC).

SECONDARY OBJECTIVES:

I. To explore the toxicity, response rate (RR) and progression free survival (PFS) in three expanded cohorts of heavily pre-treated FRalpha-positive a) TNBC patients; b) endometrial cancer patients; and c) ovarian, primary peritoneal, or fallopian tube cancer patients, all treated at the initial recommended phase II dose.

II. To provide additional safety data from the expanded cohorts to help inform on the RP2D for each cohort.

III. To evaluate the relationship between intratumoral levels of DM4, tumoral expression of FRalpha, and plasma concentration of DM4 at 48 and 72 hours following the first dose.

IV. To determine the pharmacokinetics (PK) of DM4 and gemcitabine when given in combination.

EXPLORATORY OBJECTIVE:

I. To evaluate the role of archival FRalpha expression as a substitute for the 48-72 hour (H) expression in determining intratumoral concentration of DM4.

OUTLINE: This is a dose escalation study.

Patients receive mirvetuximab soravtansine intravenously (IV) on day 1 and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Cycles repeat every 3 weeks in the absence of disease progression or unexpected toxicity.

After completion of study treatment, patients are follow up at 30 days and then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have one of the following pathologically documented recurrent tumor types with FRalpha positivity by the Ventana immunohistochemistry (IHC):

  * Ovarian, primary peritoneal, fallopian tube (with exclusion of low grade, clear cell or sarcomatoid histologies for ovarian cancer) >= 50% of tumor staining >= 2+ intensity
  * Endometrial >= 50% of tumor staining >= 2+ intensity
  * TNBC confirmed by medical history of HER2-negative (confirmed by IHC 0, 1+ regardless of fluorescence in situ hybridization [FISH] ratio; IHC 2+ with FISH ratio < 2.0 or HER2 gene copy < 6.0; FISH ratio of 0, indicating gene deletion; when positive and negative in situ hybridization controls are present); estrogen receptor (ER) negative (confirmed as ER expression =< 1% positive tumor nuclei); progesterone receptor (PR) negative (confirmed as PR expression =< 1% positive tumor nuclei): >= 25% of tumor staining >= 1+ intensity
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions >= 10 mm and short axis for nodal lesions >= 15 mm); patients with recurrent ovarian, primary peritoneal, fallopian tube cancer may have biochemical relapse only, with baseline values of CA-125 at least 2 X upper limit of normal (ULN)
* Treatment with targeted agents, immunotherapy, or hormones is allowed; patients are only eligible if they have received and failed, or have been intolerant to standard treatments known to confer clinical benefit
* Life expectancy of greater than 3 months
* Absolute neutrophil count >= 1.5 x 10^9/L, determined within 14 days of registration
* Platelets >= 100 x 10^9/L, determined within 14 days of registration
* Total bilirubin =< 1.5 x upper limit of normal (ULN), determined within 14 days of registration
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal, determined within 14 days of registration
* Alkaline phosphatase =< 2.5 X institutional upper limit of normal, determined within 14 days of registration
* Creatinine clearance >= 50 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal, determined within 14 days of registration
* Women of childbearing potential must have a negative pregnancy test at screening and must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 3 months after the last dose of IMGN853 and gemcitabine
* Patients must consent to analysis on archival tissue
* Ability to understand and the willingness to sign a written informed consent document
* Patients must have resolution of toxic effect(s) of the most recent prior chemotherapy to grade 1 or less (except alopecia)
* Cohort A: Patients with TNBC must have received no more than 4 lines of systemic cytotoxic chemotherapy; patients must have received and failed, or have been intolerant to anthracycline, taxanes, capecitabine, eribulin or other agents known to confer clinical benefit; patients are not required to fail all these agents if, in the investigator's opinion, patients would benefit from treatment on current protocol
* Cohort B: Patients with recurrent endometrial cancer may have received up to 2 lines of cytotoxic chemotherapy (adjuvant and one line for recurrent disease, or 2 lines of chemotherapy for recurrent uterine cancer in patients who did not receive adjuvant chemotherapy); patients must have received and failed, or have been intolerant to platinum agents, taxanes, liposomal doxorubicin or other agents known to confer clinical benefit; patients are not required to fail all these agents if, in the investigator's opinion, patients would benefit from treatment on current protocol
* Cohort C: Eligible patients must have received no more than 4 lines of systemic cytotoxic chemotherapy and must have disease resistant to platinum therapy (disease that progressed during or within six months of completing subsequent platinum therapy); primary platinum refractory patients are eligible providing they meet other eligibility criteria; in addition to platinum agents, patients must have received and failed, or have been intolerant to taxanes, liposomal doxorubicin or other agents known to confer clinical benefit; patients are not required to fail all these agents if, in the investigator's opinion, patients would benefit from treatment on current protocol
* Cohort C: Patients in this cohort only will require a single tumor biopsy 48-72H after the first administration of IMGN853 and gemcitabine on day 1, cycle 1 of treatment, providing it is safe/feasible and confers non-significant risk to patient

Exclusion Criteria:

* Previous treatment with gemcitabine
* Prior treatment with FR-targeting investigational agents is not allowed
* Patients who have had chemotherapy (including investigational cytotoxic chemotherapy), biologic agents (e.g., cytokines or antibodies) within 3 weeks (6 weeks for nitrosoureas or mitomycin C) before the first dose of study treatment
* Patients who have received radiation within 14 days before the first dose of study treatment
* Any other prior malignancy from which the patient has been disease free for less than 3 years, with the exception of adequately treated and basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of any site
* Patients with known brain metastases
* Serious concurrent illness or clinically-relevant active infection, including, but not limited to the following:

  * Known active hepatitis B or C
  * Known human immunodeficiency virus (HIV) infection
  * Varicella-zoster virus (shingles)
  * Cytomegalovirus infection
  * Any other known concurrent infectious disease, requiring IV antibiotics with 2 weeks of study enrollment
* Other intercurrent illness including, but not limited to symptomatic congestive heart failure and/or QT interval > 470 for females and > 450 for males, unstable angina pectoris, cardiac arrhythmia, hemorrhagic or ischemic stroke within the last 6 months or psychiatric illness/social situations that would limit compliance with study requirements
* History of interstitial pneumonitis
* History of cirrhotic liver disease
* Presence of > grade 1 peripheral neuropathy
* Active or chronic corneal disorder, including but not limited to the following: Sjogren's syndrome, Fuchs corneal dystrophy (requiring treatment), history of corneal transplantation, active herpetic keratitis, and also active ocular conditions requiring on-going treatment/monitoring such as wet age-related macular degeneration requiring intravitreal injections, active diabetic retinopathy with macular edema, presence of papilledema, and acquired monocular vision
* Major surgery within 2 months prior to enrollment or minor surgery within 7 days of the first day of treatment
* History or evidence of thrombotic or hemorrhagic disorders within 6 months before first study treatment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to gemcitabine or IMGN853
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with gemcitabine or IMGN853
* Required used of folate-containing supplements (e.g. folate deficiency)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose assessed by Common Terminology Criteria for Adverse Events version 4 | Up to 3 weeks
  Tables will be created to summarize toxicities by dose level, cycles delivered, and total dose delivered, and side effects by dose and by cycle.

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events and clinically significant >= grade 3 changes assessed by Common Terminology Criteria for Adverse Events version 4.0 | Up to 2 years
  Will assess the type, severity and attribution, time to onset, and duration.
Response | Up to 2 years
  Will be assessed by Response Evaluation Criteria in Solid Tumors 1.1.
Progression free survival | Time from study entry to disease progression, assessed up to 2 years
Assessment of biological correlatives assessed by biopsy | Up to 2 years

OTHER OUTCOMES:
FRalpha expression | Day 1
  FRalpha expression at baseline (in archival tissue) and in a single research biopsy (Cohort C only) at 48-72H will be correlated to intratumoral and circulating levels of DM4. Will develop a model incorporating both blood levels and FRalpha expression as predictors of DM4 intratumoral drug concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Edward W Wang, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - City of Hope Upland, Upland, California